CLINICAL TRIAL: NCT06384482
Title: To Evaluate the Safety and Pharmacokinetic of SNC115 Injections in Patients With Recurrent/Refractory Small Cell Lung Cancer and Lung Large Cell Neuroendocrine Crcinoma: an Open-label, Single-arm, Dose Escalation Exploratory Study
Brief Title: SNC115 Injections in Patients With Recurrent/Refractory Small Cell Lung Cancer and Lung Large Cell Neuroendocrine Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Simnova Biotechnology Co.,Ltd. (Industry)
Collaborators: Shanghai Chest Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNC115-DLL3 CART-101
Record Dates: First submitted 2024-04-10; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Recurrent/Refractory Small Cell Lung Cancer Lung Large Cell Neuroendocrine Carcinoma
Keywords: DLL3 CAR-T small cell lung cancer Lung large cell neuroendocrine carcinoma
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: SNC115 injection

INTERVENTIONS:
Drug: SNC115 injection — SNC115 Injection is DLL3 CART.

SUMMARY:
This study is a FIH dose escalation clinical study, with single arm, open label and design, in order to observe the preliminary safety and Pharmacokinetic of SNC115 Injection in participants with Recurrent/refractory small cell lung cancer and Lung large cell neuroendocrine carcinoma.

DETAILED DESCRIPTION:
The study will enroll at most 35 participants diagnosed with Recurrent/refractory small cell lung cancer or Lung large cell neuroendocrine carcinoma.

There will be about 5 preset dose groups in this clinical trial, Participants will be enrolled from low dose group to high dose group. Dose escalation will be decided by the SRC (Safety Review Committee). There will be expanded cases in the aim dose group.

The protocol will be performed into Screening period (-30+ days), Mononuclear cells acquisition, Lymphodepletion (-5~-3 days), SNC115 Injection infusion and DLT observation period (day 0~28days), and follow-up period (1-5 years). According to the administration strategy, we will start from single administration.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, regardless of gender;
2. Histological or cytological diagnosis of SCLC or pulmonary LCNEC (WHO 2021)
3. Relapse or refractory after receiving at least first-line standard therapy, or inability to tolerate first-line standard therapy
4. Eastern Cooperative Oncology Group score 0-1;
5. At least one measurable tumor lesion (other than brain metastases) according to solid tumor response criteria 1.1 (RECIST1.1)
6. Measurable lesions with an expected survival of more than 3 months;
7. Expected survival ≥12 weeks.
8. Adequate organ and bone marrow function.
9. The subjects agreed to use reliable contraceptive methods for contraception within 1 year from the signing of informed consent to reinfusion.
10. Voluntarily participate in clinical trials and sign informed consent.

Exclusion Criteria:

1. Known allergic reaction, hypersensitivity, intolerance or contraindication to SNC115 Injection or any component of drugs that may be used in the study (including fludarabine, cyclophosphamide and Tocilizumab).
2. Have received any previous CAR-T therapy or other gene-modified cell therapy.
3. Have received any previous treatment targeting DLL3.
4. Uncontrolled pleural effusion, pericardial effusion, and ascites (uncontrolled refers to repeated drainage).
5. Untreated (including new lesions or progression after previous treatment) or symptomatic brain metastases.
6. Have medical history of study excluded thrombosis, Systemic autoimmune disease, cardiopathy, cancer, infection disease and so on.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety of SNC115 Injection | Day 1 through Month 18
  Safety of SNC115 Injection will be assessed by incidence and severity of AEs and SAEs.
Safety of SNC115 Injection | Day 1 through Month 18
  Safety of SNC115 Injection will be assessed by occurrenced rate of DLT.

SECONDARY OUTCOMES:
-Efficacy of SNC115 Injection | Day 1 through Month 18
  Efficacy of SNC115 will be characterized by ORR,according to investigator assessment referring RECISIT 1.1.
-Efficacy of SNC115 Injection | Day 1 through Month 18
  Efficacy of SNC115 will be characterized by DoR,according to investigator assessment referring RECISIT 1.1.
-Efficacy of SNC115 Injection | Day 1 through Month 18
  Efficacy of SNC115 will be characterized by DCR,according to investigator assessment referring RECISIT 1.1.
-Efficacy of SNC115 Injection | Day 1 through Month 18
  Efficacy of SNC115 will be characterized by PFS,according to investigator assessment referring RECISIT 1.1.
-Efficacy of SNC115 Injection | Day 1 through Month 18
  Efficacy of SNC115 will be characterized by OS,according to investigator assessment referring RECISIT 1.1.
-Efficacy of SNC115 Injection | Day 1 through Month 18
  Efficacy of SNC115 will be characterized by TTR,according to investigator assessment referring RECISIT 1.1.

OTHER OUTCOMES:
-PK characteristic of SNC115 Injection. | Day 1 through Month 18
  PK parameters will include Cmax .
-PK characteristic of SNC115 Injection. | Day 1 through Month 18
  PK parameters will include Tmax.
PK characteristic of SNC115 Injection. | Day 1 through Month 18
  PK parameters will include AUC0-28d.
PK characteristic of SNC115 Injection. | Day 1 through Month 18
  PK parameters will include AUC0-last.
PK characteristic of SNC115 Injection. | Day 1 through Month 18
  PK parameters will include Clast.
PK characteristic of SNC115 Injection. | Day 1 through Month 18
  PK parameters will include Tlast .

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China